CLINICAL TRIAL: NCT06875544
Title: Clinical Performance of High Viscosity Bioactive Injectable Composite in Deep Marginal Elevation Randomized Controlled Trail
Brief Title: Clinical Performance of High Viscosity Bioactive Injectable Composite in Deep Marginal Elevation
Acronym: Randomized
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Sherif Hamza, Dentist, Future University in Egypt
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: Deep margin Elevation
Record Dates: First submitted 2025-03-07; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: DME; Dental; Deep Margin Elevation
Keywords: deep margin elevation
MeSH Terms: interventions — Beautifil Flow Plus F00

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bioactive injectable giomer (Active Comparator): Deep margin elevation and subsequent restoration will be done using bioactive giomer material
  Interventions: Other: Beautifil F00
- Nanohybrid injectable composite (Active Comparator)
  Interventions: Other: G-aenial Universal Injectable Flowable Composite

INTERVENTIONS:
Other: Beautifil F00 — Beautifil F00 is bioactive giomer resin composite.
  Arms: Bioactive injectable giomer
Other: G-aenial Universal Injectable Flowable Composite — Nanohybrid resin composite is a type of restorative material that features nano-sized fillers as a main component
  Arms: Nanohybrid injectable composite

SUMMARY:
Using a bioactive resin composite in subgingival Class II cavities can provide enhanced caries resistance by releasing multiple ions, including fluoride. This approach offers greater resistance to caries due to the incorporation of surface pre-reacted glass filler (S-PRG) technology (Imazato, Nakatsuka et al., 2023).

This type of composite may improve the outcomes of deep subgingival margin elevation, benefiting both restorative success and periodontal health.

ELIGIBILITY:
Inclusion Criteria:

1. Adult Patient (20-50 years old)
2. Good oral hygiene (plaque index 0 or 1)
3. Patient approval
4. Absence of parafunctional habits and/or bruxism
5. No endodontic treatment
6. No abscess
7. No partial or fixed denture

Exclusion Criteria:

1. Patients with known allergic or adverse reaction to the tested materials.
2. Bad oral hygiene
3. Systematic disease that may affect participation.
4. Xerostomic patients.
5. Patients with active periodontal disease.
6. Heavy smokers (those who smoke greater than or equal to 25 or more cigarettes a day)
7. Orthodontic treatment patient

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Recurrent caries | T (Time): T1: 1 week hours Baseline T2: 6 Months T3: 12 Months
  * 0: no evidence of caries continuous along the margin
  * 1: caries evident continuous with the margin of restoration

SECONDARY OUTCOMES:
1. Post-operative sensitivity. 2. Fracture of Restoration. 3. Bleeding on probing | T (Time): T1: 1 week hours Baseline T2: 6 Months T3: 12 Months
  1. Post-operative sensitivity.
     * 1: Absent
     * 2: Present
  2. Fracture of Restoration.
     * 1: Restoration is intact and fully retained.
     * 2: Restoration is partially retained with some portion of the restoration still intact.
     * 3: Restoration is completely missing
  3. Bleeding on probing
     * 0: Healthy gums
     * 1: Bleeding on probing 2:periodontal problem with bone loss

REFERENCES:
- [Background] Imazato S, Nakatsuka T, Kitagawa H, Sasaki JI, Yamaguchi S, Ito S, Takeuchi H, Nomura R, Nakano K. Multiple-Ion Releasing Bioactive Surface Pre-Reacted Glass-Ionomer (S-PRG) Filler: Innovative Technology for Dental Treatment and Care. J Funct Biomater. 2023 Apr 21;14(4):236. doi: 10.3390/jfb14040236. PMID 37103326
- [Background] Takatsuka T, Hirano J, Matsumoto H, Honma T. X-ray absorption fine structure analysis of the local environment of zinc in dentine treated with zinc compounds. Eur J Oral Sci. 2005 Apr;113(2):180-3. doi: 10.1111/j.1600-0722.2005.00194.x. PMID 15819827
- [Background] Yoneda M, Suzuki N, Masuo Y, Fujimoto A, Iha K, Yamada K, Iwamoto T, Hirofuji T. Effect of S-PRG Eluate on Biofilm Formation and Enzyme Activity of Oral Bacteria. Int J Dent. 2012;2012:814913. doi: 10.1155/2012/814913. Epub 2012 May 27. PMID 22693508
- [Background] Almeida Ayres AP, Tabchoury CP, Bittencourt Berger S, Yamauti M, Bovi Ambrosano GM, Giannini M. Effect of Fluoride-containing Restorative Materials on Dentin Adhesion and Demineralization of Hard Tissues Adjacent to Restorations. J Adhes Dent. 2015 Aug;17(4):337-45. doi: 10.3290/j.jad.a34555. PMID 26258176
- [Background] Basheer RR, Hasanain FA, Abuelenain DA. Evaluating flexure properties, hardness, roughness and microleakage of high-strength injectable dental composite: an in vitro study. BMC Oral Health. 2024 May 10;24(1):546. doi: 10.1186/s12903-024-04333-3. PMID 38730400
- [Background] Elderiny HM, Khallaf YS, Akah MM, Hassanein OE. Clinical Evaluation of Bioactive Injectable Resin Composite vs Conventional Nanohybrid Composite in Posterior Restorations: An 18-Month Randomized Controlled Clinical Trial. J Contemp Dent Pract. 2024 Aug 1;25(8):794-802. doi: 10.5005/jp-journals-10024-3737. PMID 39653674
- [Background] Jung JH, Park SH. Comparison of Polymerization Shrinkage, Physical Properties, and Marginal Adaptation of Flowable and Restorative Bulk Fill Resin-Based Composites. Oper Dent. 2017 Jul/Aug;42(4):375-386. doi: 10.2341/16-254-L. Epub 2017 Apr 12. PMID 28402737
- [Background] Eggmann F, Ayub JM, Conejo J, Blatz MB. Deep margin elevation-Present status and future directions. J Esthet Restor Dent. 2023 Jan;35(1):26-47. doi: 10.1111/jerd.13008. Epub 2023 Jan 5. PMID 36602272
- [Background] TY - JOUR AU - Yadav, Seema PY - 2021/11/26 SP - 20 EP - 21 T1 - DENTAL DEFECTS WITH SUBGINGIVAL EXTENSION: A RESTORATIVE CONUNDRUM VL - 10 DO - 10.36106/ijsr/9500645 JO - International Journal of Scientific Research ER -
- [Background] Eltahlah D, Lynch CD, Chadwick BL, Blum IR, Wilson NHF. An update on the reasons for placement and replacement of direct restorations. J Dent. 2018 May;72:1-7. doi: 10.1016/j.jdent.2018.03.001. Epub 2018 Mar 6. PMID 29522787
- [Background] TY - JOUR AU - Salah, Zahraa AU - Sleibi, Ahmed AU - Bissasu, Sami PY - 2024/06/30 SP - 124 EP - 137 T1 - Materials used for deep margin elevation (Review article) VL - 20 DO - 10.32828/mdj.v20i1.898 JO - Mustansiria Dental Journal ER -
- [Background] TY - JOUR AU - Magne, Pascal AU - Spreafico, R.C. PY - 2012/01/01 SP - 86 EP - 96 T1 - Deep margin elevation: A paradigm shift VL - 2 JO - Amer J Esthet Dent ER -
- [Background] Veneziani M. Adhesive restorations in the posterior area with subgingival cervical margins: new classification and differentiated treatment approach. Eur J Esthet Dent. 2010 Spring;5(1):50-76. PMID 20305873
- [Background] TY - JOUR AU - Alhumaidan, Ghaida AU - Alammar, Raghad AU - Alasmari, Dhafer AU - Alenezi, Ali PY - 2022/01/16 SP - 100034 T1 - Clinical performance of indirect restorations with cervical margin relocation in posterior teeth: A systematic review VL - 2 DO - 10.1016/j.dentre.2022.100034 JO - Dentistry Review ER -
- [Background] TY - JOUR AU - Ingamells, Hannah AU - Golenia, Katie AU - Puryer, James AU - Dorri, Mojtaba PY - 2018/01/02 SP - 24 EP - 29 T1 - Prevalence of proximal caries in adults and children at Bristol Dental Hospital and South Bristol Community Hospital VL - 9 DO - 10.1308/rcsfdj.2018.24 JO - Faculty Dental Journal ER -
- [Background] TY - CHAP AU - Anil, Aiswarya AU - Ibraheem, Wael AU - Meshni, Abdullah AU - Preethanath, Reghunathan AU - Anil, Sukumaran PY - 2022/09/26 SP - SN - 978-1-80356-359-6 T1 - Demineralization and Remineralization Dynamics and Dental Caries VL - DO - 10.5772/intechopen.105847 ER -